CLINICAL TRIAL: NCT06539026
Title: Ultrasound Assessment of Inferior Vena Cava Collapsibility Index (IVCCI) to Guide Pre-operative Fluid Management in Critically Ill Pre-eclamptic Patients in Comparison with the Standard Fluid Management
Brief Title: Inferior Vena Cava Collapsibility Index Guide for Preoperative Fluid Therapy in Preeclampsia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R146/2024
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-07

CONDITIONS: Pre-Eclampsia; Hypotension; Fluid Overload
MeSH Terms: conditions — Pre-Eclampsia; Hypotension; Edema | interventions — Fluid Therapy

STUDY DESIGN:
Intervention Model Description: a prospective, randomized, parallel-group, superior, controlled single-blinded clinical study
Who Masked: Care Provider, Outcomes Assessor
Masking Description: * The care provider intraoperative; both the anesthesiologist and the obstetrician will be blinded regarding the intervention.
  * The anesthetic residents who will assess the outcome of hypotension are blind regarding the group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IVCCI-guided fluid therapy (Experimental): the participants in this group will receive crystalloids according to the IVCCI assessment as follows:
  1. If ≥ 50 % a bolus will be given 300 ml by dripping within 30 minutes, the fluid will be repeated by half the amount if needed to reach equal or less than 40% collapsibility.
  2. If < 50 % or B line finding in lung ultrasound no bolus will be given.
  Interventions: Other: fluid therapy, 300 ml of crystalloid Ringer's solution.
- Conventional fluid therapy (No Intervention): the participants in this group will receive the standard regimen; no routine additional fluid within half an hour before surgery only the fixed maintenance of 80-100 ml/hr.

INTERVENTIONS:
Other: fluid therapy, 300 ml of crystalloid Ringer's solution. — 300 ml by dripping within 30 minutes, the fluid will be repeated by half the amount if needed to reach equal or less than 50% collapsibility.
  the fluid that will be used is sterile Ringer's solution which is an isotonic intravenous solution with pH 5.0 - 7.5 and an osmolality of 308mOsmol/kg.
  Arms: IVCCI-guided fluid therapy

SUMMARY:
The routine assessment of fluid status depends on clinical evaluation and invasive monitoring. The clinical assessment lacks objectivity and the invasive monitoring carries risks. Point of care ultrasound (POCUS) parameters can be useful as early markers of fluid status and were used in safe fluid assessment in term pregnancy and preeclampsia.

DETAILED DESCRIPTION:
Fluid therapy in preeclamptic patients presents a challenge. volume expansion may precipitate pulmonary edema while fluid restriction may worsen renal function and may aggravate post-spinal hypotension during cesarean section.

Pre-eclampsia predisposes to maternal mortality. It presents a serious hypertensive disorder during pregnancy which may progress rapidly to serious complications, including the death of both mother and fetus The optimal fluid management strategy constitutes a cornerstone in the management. The Royal College of Obstetricians and Gynecologists (RCOG) guidelines for severe pre-eclampsia recommend restrictive fluid therapy, in keeping with the absence of evidence favoring volume expansion. Restrictive management is advocated by The Society of Obstetric Medicine of Australia and New Zealand (SOMANZ) with additional fluid administration only recommended before intravenous hydralazine, regional anesthesia, immediate delivery, or in oliguric patients where a volume deficit is suspected.

Overall, limited evidence exists regarding the effectiveness of ultrasound assessment of the IVC collapsibility index to guide pre-operative fluid management in critically ill pre-eclamptic patients. A meta-analysis stated that few research trials are available in the obstetric population. Some studies suggest that it can accurately predict fluid responsiveness, but others argue that it may not be helpful.

Our trial is the first trial that compares the efficacy of IVCCI-guided perioperative fluid therapy against standard fluid therapy guided by clinical parameters in critically ill pre-eclamptic patients.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill pre-eclamptic patients for cesarean section

Exclusion Criteria:

* Patient refusal
* severe cardiovascular disease ( ejection fraction < 40 mmHg ), tricuspid regurge.
* contraindication for spinal anesthesia.
* failure to perform spinal anesthesia.
* severe hepatic.
* renal dysfunction

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2024-11-29 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
post-spinal hypotension | 20 minutes after the spinal anesthesia injection
  post-spinal anesthesia and early intraoperative (0-20 min) hypotension (MAP < 65 mmHg and/or ≥ 20% decrease from baseline. Measured by the occurrence or not of hypotension.
  The aggregation method will be according to the distribution of data if normal mean and SD will be used.

SECONDARY OUTCOMES:
occurrence of complication | from spinal anesthesia till the delivery of the fetus, or within 30 minutes postspinal which comes first
  occurrence of any complications such as pulmonary edema, need for intraoperative vasopressors.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
de-identified individual participant data (IPD) will be available to other researchers
Supporting Information: Study Protocol
Time Frame: After publishing the protocol in a relevant journal. will be available through that journal and according to the regulation
Access Criteria: the published protocol will be either free or through a subscription according to the journal.

REFERENCES:
- [Background] Chang YJ, Liu CC, Huang YT, Wu JY, Hung KC, Liu PH, Lin CH, Lin YT, Chen IW, Lan KM. Assessing the Efficacy of Inferior Vena Cava Collapsibility Index for Predicting Hypotension after Central Neuraxial Block: A Systematic Review and Meta-Analysis. Diagnostics (Basel). 2023 Aug 31;13(17):2819. doi: 10.3390/diagnostics13172819. PMID 37685357
- [Background] Gagne MP, Richebe P, Loubert C, Drolet P, Gobert Q, Denault A, Zaphiratos V. Ultrasound evaluation of inferior vena cava compression in tilted and supine term parturients. Can J Anaesth. 2021 Oct;68(10):1507-1513. doi: 10.1007/s12630-021-02051-w. Epub 2021 Jul 1. PMID 34212308
- [Background] Hernandez CA, Reed KL, Juneman EB, Cohen WR. Changes in Sonographically Measured Inferior Vena Caval Diameter in Response to Fluid Loading in Term Pregnancy. J Ultrasound Med. 2016 Feb;35(2):389-94. doi: 10.7863/ultra.15.04036. Epub 2016 Jan 18. PMID 26782160
- [Background] Pretorius T, van Rensburg G, Dyer RA, Biccard BM. The influence of fluid management on outcomes in preeclampsia: a systematic review and meta-analysis. Int J Obstet Anesth. 2018 May;34:85-95. doi: 10.1016/j.ijoa.2017.12.004. Epub 2017 Dec 20. PMID 29398426